CLINICAL TRIAL: NCT00195130
Title: Prognostic Measures in Ambulatory Care Settings
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Other Study IDs: 0397-727
Record Dates: First submitted 2005-09-15; First posted 2005-09-19 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: General Internal Medicine Patients
Keywords: prognosis; risk of death; morbidity; mortality; quality of life

INTERVENTIONS:
Behavioral: There are no interventions in this study

SUMMARY:
The primary objective of this prospective study is to develop a new method of classifying the prognosis of ambulatory patients according to their risk of long term mortality, institutionalization, morbidity (including the deterioration of pre-existing conditions or development of new problems) and functional deterioration.

DETAILED DESCRIPTION:
Specifically, from a random sample of 2000 patients taken from a cohort of established patients followed for at least three years in a general medicine practice, the objectives are:

1. to identify the demographic, clinical, and functional status variable that predict the risk of death, morbid events (e.g., the development of new complications or deterioration of existing conditions), or the deterioration in functional status using a half of the cohort chosen at random;
2. to combine these findings into a prognostic scale that can be employed in routine clinical practice; and
3. to validate the performance of this scale in the second half of the cohort.

There are no interventions in this study. Patients already under medical care by Cornell physicians will be enrolled. The only requirements for patients are to complete the questionnaires on an annual basis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are currently under the care of Physicians at Cornell Internal Medicine Associates.

Exclusion Criteria:

1. Patients who do not wish to participate in the study.
2. Patients who are not able to provide informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 1998-01; Study Completion 1999-01

PRIMARY OUTCOMES:
To develop a new method of classifying the prognosis of ambulatory patients according to their risk of long term mortality, institutionalization, morbidity and functional deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College at Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York, United States